CLINICAL TRIAL: NCT05800158
Title: Butterfly (IVD -TAQPATH V1 510K) - Clinical Performance Study Protocol - PRJ0003622
Brief Title: Butterfly - Clinical Performance Study
Status: Completed | Type: Observational
Sponsor: Thermo Fisher Scientific, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: PCP0131832
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: COVID-19; Coronavirus Infections
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasopharyngeal and anterior nasal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SARS-CoV-2: Nasopharyngeal and anterior nasal swabs collected from symptomatic individuals suspected of COVID-19 by their health care provider.
  Interventions: Diagnostic Test: Applied Biosystems™ TaqPath™ COVID-19 Diagnostic PCR Kit

INTERVENTIONS:
Diagnostic Test: Applied Biosystems™ TaqPath™ COVID-19 Diagnostic PCR Kit — A reverse transcription, real-time polymerase chain reaction (RT-qPCR) test for the qualitative detection of SARS-CoV-2.

SUMMARY:
This prospective clinical performance study is a non-interventional, multi-center study to evaluate the assay performance of the COVID-19 test using upper respiratory specimens. Prospectively collected nasopharyngeal and anterior nasal swabs will be collected from each participant recruited in the study.

DETAILED DESCRIPTION:
The Applied Biosystems™ TaqPath™ COVID-19 Diagnostic PCR Kit (referred to as "COVID-19 test") aims to develop a reverse transcription, real-time polymerase chain reaction (RT-qPCR) test for the qualitative detection of SARS-CoV-2.

The purpose of this study is to evaluate the clinical performance of the TaqPath™ COVID-19 Diagnostic PCR Kit (COVID-19 test) in nasopharyngeal swabs and anterior nasal swabs from symptomatic individuals suspected of COVID-19 by their health care provider.

A composite comparator approach will be used to evaluate the performance of the COVID-19 test which includes the use of three highly sensitive SARS-CoV-2 molecular assays as comparators. Clinical calls will be compared between COVID-19 test and the three composite comparators. The third comparator assay will only be used to test samples that show discrepant clinical calls between the first two comparator methods, for a two-out-of-three result interpretation. The Clinical Performance Study Protocol (CPS Protocol) outlines the clinical sample collection and testing protocols which will be used to satisfy the FDA 510(k) study requirements in the US.

ELIGIBILITY:
Inclusion Criteria:

Participants of all ages must meet the following inclusion criteria to be eligible for participation in the study:

* Ability to provide informed consent or assent (as age-appropriate). Stated willingness and ability to comply with the study procedures including nasopharyngeal and anterior nasal swab collection.
* Individuals with at least one of the following COVID-19 symptoms:

  1. fever or chills
  2. congestion or runny nose
  3. headache or fatigue
  4. muscle or body aches

  b. new loss of taste or smell c. a new or worsening cough or sore throat d. shortness of breath or difficulty breathing e. decrease in appetite, nausea, vomiting, diarrhea.
* Subjects suspected of having COVID-19 symptoms for seven (7) or fewer days.

Exclusion Criteria:

Participants meeting the following criterion will be excluded from the study:

* Subjects suspected of having COVID-19 symptoms for greater than seven (7) days.
* Subjects who have provided upper respiratory tract samples for other clinical studies within twenty-four (24) hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be composed of participants suspected of COVID-19. After a subject is determined eligible for study participation (met inclusion criteria and did not meet exclusion criteria) and has completed the institutional review board (IRB)-approved informed consent form process (or assent, as age appropriate), the subject is enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Clinical performance evaluation of the COVID-19 test | Between April 2023 and August 2023
  Clinical performance evaluation of the COVID-19 test using a composite comparator approach with upper respiratory specimens to meet PPA and NPA requirements.
Identification of adverse events | Between April 2023 and August 2023
  Identify any adverse events or complications associated with the COVID-19 test

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - KUR Research at Exer Urgent Care - Manhattan Beach, Manhattan Beach, California
  - KUR Research at Exer Urgent Care - Redondo Beach, Redondo Beach, California
  - Medical Center for Clinical Research, San Diego, California
  - Multi Specialty Research Associates, Lake City, Florida
  - D&H National Research Centers, Miami, Florida
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - KUR Research at AFC Urgent Care, The Bronx, New York
  - KUR Research at AFC Urgent Care, Easley, South Carolina
  - KUR Research at AFC Urgent Care, Powdersville, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - KUR Research at CityDoc Urgent Care, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No